CLINICAL TRIAL: NCT05730998
Title: The Beneficial Effects of a Cranberry-based Oral Nutritional Supplement on the Prevention of Urinary Tract Infections in Diabetic Subjects
Brief Title: Cranberry for the Prevention of Urinary Tract Infections
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Azienda di Servizi alla Persona di Pavia (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 2207/01072022
Record Dates: First submitted 2023-02-07; First posted 2023-02-16 (Actual); Last update posted 2023-02-16 (Actual); Status verified 2023-02

CONDITIONS: Diabetes; Urinary Infection
MeSH Terms: conditions — Diabetes Mellitus; Urinary Tract Infections

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): 1 capsule (120 mg) of Anthocran phytosome will be taken 1 times a day, for 6 months, with control every 2 months and phone call every month of treatment.
  Interventions: Dietary Supplement: ANTHOCRAN FITOSOMA
- Placebo group (Placebo Comparator): 1 capsule of placebo will be taken 1 times a day, for 6 months, with control every 2 months and phone call every month of treatment.
  Interventions: Dietary Supplement: PLACEBO

INTERVENTIONS:
Dietary Supplement: ANTHOCRAN FITOSOMA — The product (Anthocran phytosome or placebo) will be taken in the quantity of 1 capsule of 120 mg, 1 times a day, for 6 months
  Arms: Intervention group
Dietary Supplement: PLACEBO — Placebo will be taken in the quantity of 1 capsule of 120 mg, 1 times a day, for 6 months
  Arms: Placebo group

SUMMARY:
This research aims to evaluate the potential benefit of an oral nutritional supplement based on Anthocran phytosome compared to placebo on the prevention of urinary infections, including microbiota analyzes, in postmenopausal women (> 70 years) with diabetes.

For each subject enrolled, all parameters relating to urinary infections will be assessed at the beginning (baseline), every 2 months from the start of treatment and at the end of treatment (6 months), with urine analysis and quality of life questionnaires.

ELIGIBILITY:
Inclusion Criteria:

* postmenopausal women (> 70 years) with diabetes.
* treatment with SGLT-2 inhibitors
* disease duration for at least 10 years, with at least 1 episode of infection the previous year and Charlson's co-morbidity index> 6.

Min Age: 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 60 (Actual)
Dates: Start 2022-09-01 (Actual); Primary Completion 2022-12-31 (Actual); Study Completion 2023-01-31 (Actual)

PRIMARY OUTCOMES:
urinalysis | At baseline
  Urinalysis included color, specific gravity, pH, glucose, protein, red blood cell, white blood cell. Microscopic examinations were performed under a clinical light microscope (Olympus Opto Systems India Pvt. Ltd. New Delhi, India).
urinalysis | After two months of treatment
  Urinalysis included color, specific gravity, pH, glucose, protein, red blood cell, white blood cell. Microscopic examinations were performed under a clinical light microscope (Olympus Opto Systems India Pvt. Ltd. New Delhi, India).
urinalysis | After four months of treatment
  Urinalysis included color, specific gravity, pH, glucose, protein, red blood cell, white blood cell. Microscopic examinations were performed under a clinical light microscope (Olympus Opto Systems India Pvt. Ltd. New Delhi, India).

SECONDARY OUTCOMES:
urine culture | At baseline
  A positive urinary culture was defined as growth of a single urine pathogen of >104 cfu/mL urine specimen.
urine culture | After two months of treatment
  A positive urinary culture was defined as growth of a single urine pathogen of >104 cfu/mL urine specimen.
urine culture | After four months of treatment
  A positive urinary culture was defined as growth of a single urine pathogen of >104 cfu/mL urine specimen.
urine culture | After six months of treatment
  A positive urinary culture was defined as growth of a single urine pathogen of >104 cfu/mL urine specimen.

CONTACTS AND LOCATIONS:
Locations (1):
- l'Istituto di Riabilitazione e cura "Santa Margherita" di Pavia, Azienda di Servizi alla Persona (ASP)., Pavia, Italy